CLINICAL TRIAL: NCT05734573
Title: Effects of Family-based Treatment on Adolescent Outpatients Treated for Anorexia Nervosa in the Eating Disorder Unit of Helsinki University Hospital
Brief Title: The Effectiveness of Eating Disorder Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Svetlana Oshukova, Doctor of medicine, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 653/13/01/03/2015/1
Record Dates: First submitted 2023-01-08; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Family-based treatment — FBT is carried out by a family therapist who has received FBT training. The duration of FBT is commonly 6-12 months, in most cases comprising 10-20 sessions. At the beginning of treatment, there are weekly sessions; later in treatment, the sessions are less frequent. The patient and their family meet their psychiatrist every four to six weeks, and the family therapist also takes part in these meetings. The treatment is implemented in accordance with the FBT treatment manual.

SUMMARY:
Family-based treatment (FBT), a form of family therapy for eating disorders (ED) in young patients, has proven to be effective in numerous large-scale studies. This study aims to evaluate outcomes of the treatment for anorexia nervosa (AN) in a 'real-world' setting in a specialized outpatient clinic in Helsinki, Finland. Fifty-two young female patients seen for treatment between June 2013 and December 2017 were included in the study. Demographic and treatment characteristics, weight, and ED symptoms before and after treatment are reported

DETAILED DESCRIPTION:
Aim: The naturalistic outcome of outpatient FBT for adolescent AN was investigated.

Methods: Fifty-two female patients and their families who received FBT at a tertiary eating disorders unit participated in the study. Data on their pre-treatment parameters, treatment details, and condition at the end of treatment (EOT) was collected from their medical records

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Anorexia nervosa
* Admitted to FBT at the Eating Disorder Unit from June 1, 2013, through December 31, 2017

Exclusion Criteria:

* No exclusions

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
% of patients with body weight normalization in treatment | Treatment period, aprox. 1 year
  Rate of patients with a normal body weight defined as a BMI over 18.5 at the end of treatment was calculated.
% of patients with eating disorder symptoms at the end of treatment | Treatment period, aprox. 1 year
  The data of any eating disorder symptoms detected by a psychiatrist at the end of treatment were collected from the medical records, and the incidence was calculated.
% of patients in need for a further treatment after the intervention | Treatment period, aprox. 1 year
  Rate of patients who still needed treatment after the FBT intervention from was assessed at the end of treatment. The data were obtained from the medical files of the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jaana Suokas, Dos, Study Director — Helsinki University Central Hospital

IPD SHARING:
Plan to Share IPD: No
The dataset generated for the study is not publicly available due to privacy restrictions. The data are available on request from the principal investigator

REFERENCES:
- [Background] Jones M, Volker U, Lock J, Taylor CB, Jacobi C. Family-based early intervention for anorexia nervosa. Eur Eat Disord Rev. 2012 May;20(3):e137-43. doi: 10.1002/erv.2167. Epub 2012 Mar 22. PMID 22438094
- [Background] Lock J. Family therapy for eating disorders in youth: current confusions, advances, and new directions. Curr Opin Psychiatry. 2018 Nov;31(6):431-435. doi: 10.1097/YCO.0000000000000451. PMID 30063479
- [Background] Lock J, Le Grange D. Family-based treatment: Where are we and where should we be going to improve recovery in child and adolescent eating disorders. Int J Eat Disord. 2019 Apr;52(4):481-487. doi: 10.1002/eat.22980. Epub 2018 Dec 6. PMID 30520532
- [Derived] Oshukova S, Suokas J, Nordberg M, Algars M. Effects of family-based treatment on adolescent outpatients treated for anorexia nervosa in the Eating Disorder Unit of Helsinki University Hospital. J Eat Disord. 2023 Sep 11;11(1):154. doi: 10.1186/s40337-023-00879-9. PMID 37697396

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-21): https://cdn.clinicaltrials.gov/large-docs/73/NCT05734573/Prot_SAP_000.pdf